CLINICAL TRIAL: NCT03623581
Title: An Open-label, Single-arm, Phase II Clinical Study of Anti-PD-1 Antibody GB226 in Treatment of Relapsed/Metastatic/Unresectable Alveolar Soft Part Sarcoma (ASPS)
Brief Title: Clinical Trial in Chinese Patients of Elapsed/Metastatic/Unresectable Alveolar Soft Part Sarcoma(GB226)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gxplore-005
Record Dates: First submitted 2018-07-26; First posted 2018-08-09 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Alveolar Soft Part Sarcoma
Keywords: ASPS
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB226 3mg/kg every 2 weeks (Experimental): Geptanolimab Injection, 3mg/kg every 2 weeks
  Interventions: Biological: GB226

INTERVENTIONS:
Biological: GB226 — 3mg/kg treat every 2 weeks
  Other Names: Recombinant humanized anti-PD-1 monoclonal antibody injection; Geptanolimab

SUMMARY:
This study is a single-arm, phase 2 trial of Geptanolimab in patients with initially unresectable, recurrent or metastatic ASPS. The study aims to study the activity of Geptanolimab assessed per RECIST 1.1 and iRECIST criteria, and safety profile.

DETAILED DESCRIPTION:
Patients received Geptanolimab 3mg/kg via intraveneous infusion every 2 weeks until disease progression, death, unacceptable toxicity, withdrawal of consent or end the the study (i.e. a maximum treatment duration of one years of the last subject, termination of treatment, consent withdrawal, lost to follow-up or death, whichever occurs first).

During the treatment period, subjects were evaluated for safety (once every 2 weeks) and efficacy (once every 6 weeks)，If clinical symptoms suggestive of PD occur, an external visit should be arranged to complete the imaging evaluation and confirmation.

Geptanolimab treatment was permitted to continue beyond the first RECIST-defined progressive disease (PD), if clinical benefit was noted and the toxicity was acceptable. No dose modification was allowed, but dose discontinuation was permitted for up to six weeks for adverse events.

Safety was monitored until 30 days and/or 90 days (without initiation of another anticancer treatment) after the last dose of the study drug, for all patients received at least one dose of treatment.

At the end of the treatment, for the subjects who have not yet developed PD and have not started the subsequent anti-tumor treatment, the efficacy evaluation will continue every 6 weeks (± 7 days) in the first 3 months, and every 12 weeks thereafter, until the end of the study or withdrawal of informed consent or occurrence of PD, initiation of a new anti-tumor treatment, death or lost to follow-up.

All subjects who had received GB226 treatment at least once were required to have survival follow-up visits, which were planned every 3 months (± 14 days) after the safety follow-up / disease progression follow-up visit.

The end of the study was defined as the death, loss of visit, withdrawal of informed consent and completion of the final study visit of the last subject, and the end of treatment of the last subject for one year or the early end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion criteria:

The subjects can be enrolled only all the following criteria are met:

1. Sign the informed consent form;
2. Aged 18~75 years old, males or females;
3. ECOG score of 0-1;
4. The expected survival is 3 months or longer;
5. Histologically or cytologically confirmed relapsed or metastatic or unresectable alveolar soft part sarcoma (ASPS);
6. There is at least one measurable lesion, which is defined as lesion accurately measured in one dimension (RECIST1.1: the longest diameter of non-lymph node lesions≥10mm, the shortest diameter of lymph node lesions ≥15mm);
7. The previous treatment is completed ≥4 weeks or ≥5 half-lives of the previous therapeutic agents (whichever is shorter) before administration (at least 1 week interval between previous treatment and study enrollment); washout with nitrosoureas, mitomycin C, RANKL inhibitor for at least 6 weeks; previous radiotherapy must be performed at least 4 weeks ago; the previous monoclonal antibody treatment must be performed at least 6 weeks ago;
8. If the patients received more than 350mg/m2 cumulative dose of adriamycin, echocardiography should be performed and left ventricular ejection fraction (LVEF) ≥50%;
9. Absolute neutrophil count ≥1.5×109/L, platelet ≥100×109/L, hemoglobin (Hb) ≥80g/L;
10. Total bilirubin ≤1.5xULN (≤3xULN is allowed for known Gilbert disease), AST/ALT≤3xULN (AST and/or ALT≤5xULN is allowed for patients with hepatic metastasis), ALP≤2.5xULN (≤5xULN is allowed for patients with hepatic metastasis or bone metastasis);
11. The creatinine clearance ≥ 50mL/min/1.73m2 (calculated based on Cockcroft-Gault formula) or Cr≤1.5xULN;
12. Female subjects who are confirmed not pregnant within 72 hours before administration; female and male patients of child-bearing potential should agree to adopt adequate contraceptive methods before enrollment, during study period and 6 months after the last dose;
13. Lactating women should agree to stop breastfeeding during the study period;
14. Agree to provide archived tumor tissue specimens or fresh tissue specimens;

Exclusion criteria:

The subjects cannot be enrolled should any of or several conditions occur:

1. Subjects who received anti-PD-1 or anti-PD-L1 monoclonal antibody or targeted drugs of relevant pathways;
2. Subjects who are known to be allergic to PD-1 monoclonal antibody or any of its excipients, or subjects who are known to have medical history of allergic diseases or serious allergic constitution;
3. Subjects who received CTLA-4 antibody;
4. Subjects who have other malignant tumor diseases other than tumor treated in this study, excluding cured malignant tumors which did not relapse within 3 years before enrollment, completely resected basal cell and squamous cell skin cancer, any type of in situ carcinoma which is completely resected;
5. Active central nervous system (CNS) metastasis (regardless of whether any treatment is received), including symptomatic brain metastasis or meningeal metastasis or spinal cord compression etc.; excluding asymptomatic brain metastasis (no progression within at least 4 weeks after radiotherapy and/or no neurological symptom or sign after surgical resection, treatment with dexamethasone or mannitol is not necessary);
6. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage;
7. The toxicity of previous treatment still > grade 1 (CTCAEV4.03 criteria), excluding alopecia and neurotoxicity;
8. Subjects who have history of psychiatric disorders;
9. Subjects who have medical history of drug addiction or drug abuse;
10. Subjects with medical history of idiopathic pulmonary fibrosis or idiopathic pneumonitis, or patients who previously received radiotherapy for large size of lungs;
11. Patients with complications requiring treatment with immunosuppressive drugs or systemic or local corticosteroids at the immunosuppressive doses (prednisone > 10mg/day or equivalent dose of similar agents);
12. Medical history of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory gastrointestinal disorders, Hashimoto's thyroiditis etc. The following should be excluded: type I diabetes mellitus, hypothyroidism which can be controlled by hormone replacement therapies only, skin diseases requiring no systemic treatment (e.g., vitiligo, psoriasis), controlled celiac disease, or diseases which may not occur without stimulating factors;
13. Subjects who previously or currently have active tuberculosis;
14. Subjects with active infection requiring systemic treatment;
15. Uncontrolled hypertension (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) or pulmonary arterial hypertension or unstable angina pectoris; previous presence of myocardial infarction or received bypass grafting or stent surgery within 6 months before administration; medical history of chronic heart failure NYHA (New York Heart Association) class 3-4; Clinically significant valvular heart diseases; subjects with serious arrhythmia requiring treatment (excluding atrial fibrillation, paroxysmal supraventricular tachycardia), including QTc interval ≥450ms for males and ≥470ms for females (calculated based on Fridericia formula); cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration;
16. Subjects with complicated serious internal diseases, including but not limited to, uncontrolled diabetes mellitus, active gastrointestinal ulcer, active bleeding etc.;
17. Positive Anti-HIV, TP-Ab, HCV-Ab; positive HBV-Ag and the copies of HBV DNA are higher than the upper limit of normal of the test units;
18. Abnormal thyroid function test (TSH, FT3, FT4);
19. Expected major surgery within 28 days before administration or during treatment period;
20. It is expected that live vaccines or attenuated vaccines are given 4 weeks before administration, during treatment period or within 5 months after the last dose;
21. Subjects who participated in another clinical trial and were treated with investigational products within 30 days before screening;
22. Patients who require RANKL inhibitor (e.g., denosumab);
23. Patients who have insufficient communication, understanding and cooperation; or patients who have poor compliance and cannot guarantee to strictly follow the study protocol;
24. Subjects who are considered unsuitable for participating in this clinical study for any other reasons at the discretion of the investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by objective response rate in patients with ASPS.

SECONDARY OUTCOMES:
Progression-free survival, PFS | up to 52 weeks
  To evaluate the efficacy of GB226 as defined by progression-free survival in patients with ASPS.
Duration of response, DOR | up to 52 weeks
  To evaluate the duration of response (DOR) of GB226 in patients with ASPS.
Disease Control Rate，DCR | up to 52 weeks
  To evaluate the disease Control Rate (DCR) of GB226 in patients with ASPS.
Overall survival, OS | up to 52 weeks
  To evaluate the duration from the first administration to death because of any reason in patients with ASPS.
Incidence and severity of adverse events | up to 52 weeks
  Incidence and severity of adverse events
Incidence and severity of immune-related adverse events | up to 52 weeks
  Incidence and severity of immune-related adverse events
Incidence and severity of serious adverse events | up to 52 weeks
  Incidence and severity of serious adverse events
iORR | up to 52 weeks
  iORR
iDCR | up to 52 weeks
  iDCR
iPFS | up to 52 weeks
  iPFS
iDOR | up to 52 weeks
  iDOR
The concentration of Antidrug antibody | up to 52 weeks
  To evaluate the immunogenicity in patients with ASPS.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Doctor, Principal Investigator — Study Principal Investigator Cancer Hospital Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.